CLINICAL TRIAL: NCT04726124
Title: A Prospective, Multicenter, Randomized, Controlled Clinical Trial to Validate the Safety and Efficacy of Microwave Versus Laser Ablation of the Great Saphenous Vein in Patients With Varicose Veins
Brief Title: MicrOwave and laSer ablaTion Study (MOST Study)
Acronym: MOST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SD-LC-001
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2021-10

CONDITIONS: Varicose Veins of Lower Limb
Keywords: endovenous microwave therapy（EMT）; endovenous laser treatment（EVLT）; great saphenous vein

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Microwave Ablation Therapeutic Apparatus. Patients with primary lower extremity varicose veins were treated with endovenous microwave therapy using Microwave Ablation Therapy Apparatus. Ultrasound examination and questionnaire survey（AVVQ and VCSS) were performed at 1 week, 3 months, 6 months,12 months after treatment,drug use and adverse events were recorded to assess complications and target lesion closure rate.
  Interventions: Device: Microwave Ablation Therapeutic Apparatus
- control group (Experimental): Semiconductor Laser Treatment Apparatus. Patients with primary lower extremity varicose veins were treated with endovenous laser treatment using Semiconductor Laser Treatment Apparatus. Ultrasound examination and questionnaire survey（AVVQ and VCSS) were performed at 1 week, 3 months, 6 months, 12 months after treatment,drug use and adverse events were recorded to assess complications and target lesion closure rate.
  Interventions: Device: Microwave Ablation Therapeutic Apparatus

INTERVENTIONS:
Device: Microwave Ablation Therapeutic Apparatus — The selected and qualified subjects with primary lower extremity varicose veins were randomly treated with microwave ablation equipment or laser treatment equipment. Subjects in the two groups were returned to the hospital for follow-up at 7 days, 3 months, 6 months, 12 months after surgery, respectively, for ultrasound examination and questionnaire evaluation, medication status and adverse events were recorded, and target lesion closure rate and subject satisfaction were evaluated.
  Other Names: Semiconductor Laser Treatment Apparatus

SUMMARY:
To validate the safety and efficacy of microwave versus laser ablation of the great saphenous vein in patients with varicose veins of lower extremities

DETAILED DESCRIPTION:
A prospective, multicenter, randomized, controlled clinical trial to validate the safety and efficacy of microwave versus laser ablation of the great saphenous vein in patients with varicose veins of lower extremities

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, not older than 80 years, male or female
2. Patients clinically diagnosed as primary great saphenous vein insufficiency with reflux lasting > 0.5 seconds on duplex ultrasound
3. Patients with CEAP grade C2-C6
4. Patients who voluntarily participate in this trial, understand all the risks and benefits described in the informed consent document, and sign the written informed consent form

Exclusion Criteria:

1. Patients with diameter of target lesion vein < 2 mm or > 15 mm
2. Patients with previous surgical treatment on the target lesion or patients with acute thrombosis
3. Patients with deep vein thrombosis and superficial vein thrombosis
4. Patients with acute systemic infectious diseases
5. Patients with severe liver and kidney dysfunction (ALT > 3 times the upper limit of normal value; creatinine > 225 umol /L)
6. Patients with known uncorrectable bleeding or severe coagulopathy
7. Patients with anesthesia contraindications
8. Patients with poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg) and diabetes mellitus (fasting glucose ≥ 10.0 mmol / L)
9. Patients with non-primary varicose veins caused by post-deep vein thrombosis syndrome, KT syndrome (Klippel-Trenaunay syndrome), arteriovenous fistula, etc.
10. Patients with other diseases that may cause difficulty in conducting the trial or evaluation, such as mental illness, AIDS, malignant tumors, liver disease, cardiac insufficiency, etc. or patients whose life expectancy is less than 1 year
11. Pregnant, lactating women, or those planning on becoming pregnant during the trial
12. Patients who have participated in clinical trials of other drugs or medical devices in the past 3 months
13. Patients considered unsuitable for inclusion by investigators for other reasons

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-09-28 (Estimated); Study Completion 2022-09-28 (Estimated)

PRIMARY OUTCOMES:
the complete closure rate of great saphenous vein at 6 months after surgery | 6 months after surgery
  Complete closure: Doppler ultrasonography showed that the target vein segment of the entire treatment is closed, with no discontinuous unclosed segment more than 5 cm.
  Calculation method: Complete closure rate = number of subjects with complete closure of target vein in the group/total number of subjects in the same group × 100%.
  The B-ultrasound check is performed on subjects 6 months after the surgery for whether the target vein is completely closed, the result is recorded. After the trial is completed, the number of subjects whose target vein is completely closed is counted, and the complete closure rate of great saphenous vein is calculated.

SECONDARY OUTCOMES:
the complete closure rate of great saphenous vein at 12 months after surgery | 12 months after surgery
  Complete closure: Doppler ultrasonography showed that the target vein segment of the entire treatment is closed, with no discontinuous unclosed segment more than 5 cm.
  Calculation method: Complete closure rate = number of subjects with complete closure of target vein in the group/total number of subjects in the same group × 100%.
  The B-ultrasound check is performed on subjects 12 months after the surgery for whether the target vein is completely closed, the result is recorded. After the trial is completed, the number of subjects whose target vein is completely closed is counted, and the complete closure rate of great saphenous vein is calculated.
surgical success rate | immediately after surgery
  Successful surgery: Doppler ultrasound examination shows that the target lesion segment is closed immediately after operation.
  Calculation method: Surgical success rate = number of subjects successfully operated in this group/total number of subjects in this group × 100%
device performance evaluation | during or after surgery
  During or after the surgery, the manipulation performance of the device is evaluated by the investigator，which is include flexibility, passability, ease of use, accuracy, stability etc.. Only the device in the test group is evaluated.
changes of venous clinical severity score (VCSS) before and after treatment | screening period, 30days, 3 months, 6months, 12 months after surgery
  VCSS is performed in the screening period, 30 days after surgery, 3 months and 6 months after surgery. The VCSS includes 10 items, namely, pain, varicose veins, edema, skin pigmentation, inflammation, skin induration, number of active ulcers, ulcer size, duration of ulcers and application of compression therapy. Each item is scored from 0 to 3 according to the severity of the disease, with a total score of 30. The higher the score, the more serious the condition.
changes of Aberdeen Varicose Vein Questionnaire (AVVQ) score before and after treatment | screening period, 30 days, 3 months, 6 months, 12 months after surgery
  Aberdeen Varicose Vein Questionnaire (AVVQ) score before and after treatment AVVQ score is performed in the screening period, 30 days after surgery, 3 months and 6 months after surgery. AVVQ includes the scope of varicose veins, the degree of pain, edema, itching, pigmentation, rash and ulcers, the use of painkillers and elastic stockings, the psychological worries, and the influence of varicose veins on daily clothing, work, life and sports. Each item is scored from 0 to 3 according to the severity of the disease. The lower the score, the better the quality of life.
time of surgery | immediately after surgery
  After the surgery, the operation time is recorded. The operation time is defined as the time from the entry of the investigational device into the vein to the withdrawal of the vein after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: weiwei Wu, M.D., Principal Investigator — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hosipital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li Y, Wu W, Li Y, Li J, Sun M. Efficacy and safety of endovenous microwave ablation versus laser ablation for great saphenous vein varicosis: study protocol for a multicentre, randomised controlled non-inferiority trial. BMJ Open. 2022 May 25;12(5):e059213. doi: 10.1136/bmjopen-2021-059213. PMID 35613801